CLINICAL TRIAL: NCT07181837
Title: A Multi-Center, Open-label, Phase 1/2 Trial of the Safety and Efficacy of MVX-220 Gene Therapy Administered by Intra-Cisterna Magna Injection to Participants With Angelman Syndrome
Brief Title: A Phase 1/2 Study of the Safety and Efficacy of MVX-220 in Angelman Syndrome
Acronym: ASCEND-AS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MavriX Bio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVX-AAV-101
Record Dates: First submitted 2025-09-06; First posted 2025-09-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Angelman Syndrome
Keywords: Angelman syndrome; gene therapy; AAV; cisterna magna
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Adults ages 18-50 (Experimental): MVX-220, single dose intra cisterna magna injection
  Interventions: Genetic: MVX-220
- Cohort 2: Children ages 4-8 (Experimental): MVX-220, single dose intra cisterna magna injection
  Interventions: Genetic: MVX-220
- Cohort 3: Optional cohort, adults and children ages 4-50 (Experimental): MVX-220, single dose intra cisterna magna injection
  Interventions: Genetic: MVX-220

INTERVENTIONS:
Genetic: MVX-220 — AAVhu68 viral vector

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MVX-220 gene therapy in children and adults with Angelman syndrome with UBE3A gene deletion, uniparental disomy, or imprinting center defect genotypes.

DETAILED DESCRIPTION:
MVX-220 is an investigational gene replacement therapy intended to provide a functional copy of the UBE3A gene to individuals with Angelman syndrome. This study is designed to evaluate the safety, tolerability and efficacy of MVX-220 in participants with Angelman syndrome who have deletion, uniparental disomy, or imprinting center disorder genotypes. The study has 2 primary cohorts: Cohort 1 that includes adults followed by Cohort 2 that includes children. All patients will receive a single dose of MVX-220 administered by injection into the cisterna magna. There is no control group and all individuals will receive the gene therapy. An independent data safety monitoring board will review the safety information from Cohort 1 before individuals can be enrolled in Cohort 2. An optional cohort of adults and/or children (Cohort 3) may be enrolled based on a review of data from Cohorts 1 and 2. All patients will be required to take steroids before and for a brief period during the study to help mitigate the risk of immune response to the gene therapy. Patients will be followed for safety and efficacy for an initial 2-year period post-treatment and then transition to less frequent monitoring schedule for an additional 3 years. The total duration of follow up in the study is 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant's parent/legal guardian must provide written informed consent.
2. Symptoms consistent with AS and documented genetic confirmation of one of the following genotypes resulting in a diagnosis of AS:

   1. Full maternal UBE3A gene deletion causing AS in the region of 15q11.2-q13
   2. Uniparental disomy
   3. Imprinting center defect
3. The participant must be 18 to 50 years of age, inclusive (for adult participants), or 4 to 8 years of age, inclusive (for pediatric participants), at Screening.
4. The participant must have the ability to ambulate independently.
5. The participant must be on stable antiepileptic medications (with no changes within 1 month prior to the Screening visit, except for weight associated dose adjustments).

Key Exclusion Criteria:

1. Clinically significant medical finding other than AS, that, in the judgment of the Investigator would make the participant unsuitable for participation.
2. Laboratory abnormalities including but not limited to:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN)
   2. Total and/or fractionated bilirubin (direct and/or indirect) > ULN
   3. Gamma-glutamyl transferase (GGT) > ULN
   4. Estimated glomerular filtration rate (eGFR) below the lower limit of normal (LLN) for age
   5. Hemoglobin < 8 g/dL
   6. White blood cell (WBC) count outside the normal range for age
   7. Platelet count < LLN
   8. Partial thromboplastin time (PTT) outside the reference range
   9. PT/International normalized ratio (INR) outside the reference range
3. Any known history and/or family history of hemophagocytic lymphohistiocytosis (HLH)/macrophage activation syndrome (MAS) or multisystem inflammatory syndrome (MIS).
4. Any known history and/or family history of disordered complement function and/or complement gene mutation(s).
5. History of systemic lupus erythematous, Still's disease, rheumatoid arthritis, and/or other severe autoimmune conditions per judgment of the Investigator.
6. Any known history of thrombotic microangiopathy (TMA)/microangiopathic hemolytic anemia, or hypercoagulable conditions including, but not limited to, disseminated intravascular coagulation (DIC), deep venous thrombosis, and pulmonary embolism.
7. Current therapy with high dose immunosuppressants.
8. Prior or current treatment with an investigational drug within 6 months or 5-half-lives of the hospital admission whichever is longer.
9. Prior treatment with an antisense oligonucleotide within 1 year of hospital admission.
10. A history of gene therapy administration.
11. Any contraindication to ICM administration procedure, including contraindications to imaging, contrast use, anesthesia, or any condition that would increase the risk of adverse outcomes from the ICM procedure.
12. Any contraindication to glucocorticoid use

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest as assessed through clinical safety, laboratory tests, ECG, vital sign measurements, and physical examinations | Up to Week 104

SECONDARY OUTCOMES:
Change in communication ability as assessed by the Observer Reported Communication Ability (ORCA) measure | From Baseline to Week 104
  The ORCA measure is a caregiver reporter assessment of communication ability that was developed specifically for Angelman syndrome. The ORCA measure produces a single score that is an estimate of an individual's overall level of communication ability, with higher T-scores reflecting greater communication ability.
Change in developmental milestones as assessed by the Bayley Scale of Infant and Toddler Development, Fourth Edition (Bayley-4) | From Baseline to Week 104
  The Bayley-4 is a performance-based assessment of developmental functioning across communication, cognition, and motor skills. The total raw score reflects the sum of all the item scores within a subdomain, with higher scores reflecting greater ability.
Change in adaptive behaviors as assessed by Vineland Adaptive Behavior Scale (VABS-3) | From Baseline to Week 104
  The VABS-3 assesses adaptive behaviors across multiple domains through a clinician-directed interview of a caregiver of an individual with AS. The total raw score reflects the sum of all the item scores within a subdomain, with higher scores reflecting greater ability.
Change in Symptoms by the Angelman Severity Assessment (ASA) | From Baseline to Week 104
  The ASA is a clinician-reported outcome measure for Angelman syndrome. The clinicians rate their overall impression of the improvement in disease-related symptoms utilizing a 7-point scale, ranging from "very much improved" to "very much worse".
Change in behaviors as assessed by the Aberrant Behavior Checklist-Community (ABC-C) | From Baseline to Week 104
  The ABC-C is a caregiver-rated questionnaire that evaluates key domains in behavior. Items are assessed on a 4 point scale ranging from "not at all a problem" to "the behavior is a severe problem".
Change in ambulatory ability as assessed by the wearable device (Syde®) | From Baseline to Week 104
  The Syde is a wearable device that collects continuous data on the ambulatory ability of participants with AS.
Change in sleep parameters as assessed by a sleep diary | From Baseline to Week 104
  The sleep diary is a caregiver-reported measure of sleep in individuals with AS.
Change in health-related quality of life as assessed by Quality of Life Inventory-Disability (QI-Disability) | Baseline to Week 104
  The QI-Disability is a caregiver-reported outcome assessment of the health-related quality of life for children and adolescents with intellectual disabilities. Item are rated on a 5-point scale, ranging from "never" to "always ".
Change in viral deoxyribonucleic acid (vDNA) levels in CSF and blood | Baseline to Week 104
Change in viral DNA levels in urine and feces | From Baseline to Week 104
Change in relevant Electroencephalogram (EEG) parameters (delta power, epileptiform activity) | From Baselien through Week 104

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No